CLINICAL TRIAL: NCT02165163
Title: Virtual Reality-Based Exercise in Cancer Patients With Chemotherapy Induced Peripheral Neuropathy
Brief Title: Virtual Reality-Based Exercise in Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: iCAMP_123
Record Dates: First submitted 2014-06-13; First posted 2014-06-17 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Distorted; Balance; Motor Deficit
MeSH Terms: conditions — Neurologic Manifestations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Balance Training (Experimental): Balance training will be conducted individually two times per week for 4 weeks. Each training session will include virtual reality tasks such as "ankle reaching" and "obstacle crossing" using a virtual obstacle shown on a computer screen. Each session will last 30 - 45 minutes.
  Interventions: Other: Balance Training
- Control (No Intervention): The control group will keep their normal activity without receiving any intervention.

INTERVENTIONS:
Other: Balance Training — Balance training will be conducted individually two times per week for 4 weeks. Each training session will include virtual reality tasks such as "ankle reaching" and "obstacle crossing" using a virtual obstacle shown on a computer screen. Each session will last 30 - 45 minutes.
  Arms: Balance Training

SUMMARY:
The aim of the present study is to evaluate an innovative virtual reality-based balance training intervention for improving clinically relevant motor performances (balance and gait) in cancer patients.

The investigators hypothesize that the virtual reality-based balance training intervention will improve balance and gait performances in cancer patients compared to a control group receiving usual care only.

ELIGIBILITY:
Inclusion Criteria:

* ability to ambulate without assistance
* willingness to provide informed consent
* cancer
* neuropathy related to chemotherapy

Exclusion Criteria:

* severe neurologic, cardiovascular, metabolic, or psychiatric disorders
* severe visual impairment
* cognitive impairment

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-09; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Postural Balance | after 4 weeks
  Postural Balance during quiet standing for 30 seconds will be assessed using validated wearable sensor technologies (BalanSens™)

SECONDARY OUTCOMES:
Gait performance | 4 weeks
  Gait performance will be measured using validated wearable sensor technology (LEGSys™)

CONTACTS AND LOCATIONS:
Overall Officials: Bijan Najafi, PhD, Principal Investigator — interdisciplinary Consortium on Advanced Motion Performance (iCAMP), Department of Surgery, College of Medicine, University of Arizona
Locations (1):
- University of Arizona Cancer Center, Tucson, Arizona, United States